CLINICAL TRIAL: NCT01937533
Title: Diffusion-weighted MRI at 3T Using an Endovaginal Coil: Evaluating the Prognostic Value of the Apparent Diffusion Coefficient Distribution in Stage 1 Cervical Tumours
Brief Title: Apparent Diffusion Coefficient as a Prognostic Biomarker in Cervical Cancer
Status: Completed | Type: Observational
Sponsor: Institute of Cancer Research, United Kingdom (Other)
Collaborators: Cancer Research UK (Other)
Responsible Party: Principal Investigator, Nandita deSouza, Professor of Translational Imaging, Institute of Cancer Research, United Kingdom
Other Study IDs: 13/EE/0198 CCR3938
Record Dates: First submitted 2013-08-29; First posted 2013-09-09 (Estimated); Last update posted 2020-01-28 (Actual); Status verified 2020-01

CONDITIONS: Cancer
Keywords: Magnetic Resonance Imaging
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cervical Cancer: Patients with presumed early cervical cancer being considered for curative surgery
  Interventions: Procedure: Magnetic Resonance Imaging using an endovaginal receiver coil

INTERVENTIONS:
Procedure: Magnetic Resonance Imaging using an endovaginal receiver coil

SUMMARY:
This study aims to develop the technique of Diffusion-Weighted Magnetic Resonance Imaging(DW-MRI)for the assessment of stage 1 cervical cancers. An endovaginal receiver coil has been designed and developed at the Institute of Cancer Research and Royal Marsden NHS Foundation Trust for use at high field strengths(3T). This will be used to evaluate if DW-MRI at 3T can be used to differentiate different histological characteristics within whole tumours and so determine if the technique could be of prognostic value.

The study hypothesis is that this technique will be able to differentiate tumours with histological features known to be associated with poor prognosis (tumour type, grade and lymphovascular space invasion).

ELIGIBILITY:
Inclusion Criteria:

* All patients with presumed early stage cervical cancer being considered for curative surgery

Exclusion Criteria:

* Ferromagnetic metal implants
* claustrophobia (MRI incompatibility)

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary Care Clinic
Sampling Method: Probability Sample
Enrollment: 236 (Actual)
Dates: Start 2013-10-02 (Actual); Primary Completion 2019-05 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
To obtain histogram metrics(centiles, skew, kurtosis, entropy) for cervical cancer and compare them between histologically poor prognosis and good prognosis groups. | 1-2 months post imaging
  Pixel by pixel analysis of ADC from tumour regions of interest will be used to derive histograms and the 10th, 25th, 50th, 75th and 90th centile values and histogram skew, kurtosis and entropy values for each tumour will be recorded. The number of regions will vary with tumour volume in each patient, given the mean size of lesions in patients studied in a pilot set, it is envisaged that we will analyse 1-5 regions of interest in each tumour. The data will be analysed separately by 2 observers who will be blinded to the histopathological characteristics and assuming good inter-observer agreement, an average of their results will be used for data analysis. The difference in mean centile ADC values of the distribution and the skewness, kurtosis and entropy values between squamous vs. adenocarcinoma, well/moderately differentiated vs. poorly differentiated tumour regions and the absence vs. the presence of lymphovascular space invasion in that region will be determined.

SECONDARY OUTCOMES:
Establish ADC values associated with poor prognosis tumours | Duration of study, 2-3 years
  The centile measures of the ADC values will be summarised using means and standard deviations if the data are normally distributed and medians and ranges if the data are non-normally distributed. The unpaired t-test will be used to analyse normally distributed data and the Mann Whitney U test for non-parametric data. Point estimates for the differences between centile ADC values and other summary measures for tumour type, grade and presence or absence of lymphovascular space invasion will be derived and 95% confidence intervals attached where appropriate. The Bonferroni correction method will be used to adjust significance levels for multiple comparisons.
  The key clinical question is whether or not the imaging can differentiate poor prognosis tumours from good prognosis ones from the histogram metrics.

CONTACTS AND LOCATIONS:
Overall Officials: Nandita deSouza, Professor, Principal Investigator — ICR
Locations (1):
- The Institute of Cancer Research and Royal Marsden NHS Foundation Trust, Sutton, Surrey, United Kingdom